CLINICAL TRIAL: NCT03650946
Title: Clinical Application of 68Ga-PSMA PET in Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201508052MIND
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Ga-68 PSMA PET
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: men with high or intermediate risk localized disease who are about to undergo definitive surgery or radiotherapy
  Interventions: Diagnostic Test: Ga-68 PSMA PET
- 2: men with rising PSA after local definitive treatments
  Interventions: Diagnostic Test: Ga-68 PSMA PET
- 3: m0CRPC with a PSA >1.0 or 2.0
  Interventions: Diagnostic Test: Ga-68 PSMA PET

INTERVENTIONS:
Diagnostic Test: Ga-68 PSMA PET — Ga-68 PSMA PET

SUMMARY:
Prostate cancer is the 7th leading cause of cancer death for men in Taiwan. It is important to identify the extent of disease extent to deliver adequate treatment, either for primary staging or in recurrence. However, conventional imaging techniques including computed tomography, bone scintigraphy, and immunoscintigraphy with 111In-capromab pendetide are not sensitive or specific enough to detect metastatic or recurrent disease. Although more widely applied, magnetic resonance still relies on size and shape criteria. 68Ga-PSMA is a new novel positron emission radiotracer which several preliminary data has shown to be effective of detecting recurrent or metastatic prostate cancer. These studies are confined to a small retrospective European population. In this study we aim to synthesize the novel tracer, find the usefulness of 68Ga-PSMA PET in detecting prostate cancer, including primary staging and recurrence, explore the relationship between imaging and clinical parameters, and seek the possibility of 68Ga-PSMA PET to predict tumor nature and prognosis.

DETAILED DESCRIPTION:
Prostate cancer is the 7th leading cause of cancer death for men in Taiwan. It is important to identify the extent of disease extent to deliver adequate treatment, either for primary staging or in recurrence. However, conventional imaging techniques including computed tomography, bone scintigraphy, and immunoscintigraphy with 111In-capromab pendetide are not sensitive or specific enough to detect metastatic or recurrent disease. Although more widely applied, magnetic resonance still relies on size and shape criteria. 68Ga-PSMA is a new novel positron emission radiotracer which several preliminary data has shown to be effective of detecting recurrent or metastatic prostate cancer. These studies are confined to a small retrospective European population. In this study we aim to synthesize the novel tracer, find the usefulness of 68Ga-PSMA PET in detecting prostate cancer, including primary staging and recurrence, explore the relationship between imaging and clinical parameters, and seek the possibility of 68Ga-PSMA PET to predict tumor nature and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer

Exclusion Criteria:

* Patients with known malignancy in other organs.
* Patients with severe claustrophobia or unstable vital sigh
* Other serious comorbidities evaluated by primary investigator

Ages: 40 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 1 year
  initial staging compared to pathology, clinical and follow-up result

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan